CLINICAL TRIAL: NCT01951222
Title: Bronchodilator Properties and Safety of a Repeated Dose of V0162 in Asthma.
Brief Title: Bronchodilator Properties and Safety in Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-002517-35
Record Dates: First submitted 2013-09-05; First posted 2013-09-26 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Asthma
Keywords: Asthma, COPD, broncodilator, airway, lung, inhalation, antimuscarinic
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- V0162 dose1 (Experimental)
  Interventions: Drug: V0162
- V0162 dose2 (Experimental)
  Interventions: Drug: V0162
- placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: V0162
  Arms: V0162 dose1; V0162 dose2
Other: Placebo
  Arms: placebo

SUMMARY:
Recent large clinical studies have demonstrated the interest of LAMA therapy in the management of asthma, when compared to LABA.

V0162 is a compound with a very long lasting bronchodilator effect when compared to reference treatment in non-clinical models and in COPD patients. Secondary properties of V0162 (i.e.H1/H4 and PDE IV-inhibition) could enhance the efficacy of this antimuscarinic compound and could bring option in the treatment obstructive lung disease. The objective of the study is to assess the bronchodilator properties of V0162 during 8 days in adult patients with asthma usually treated with ICS and LABA. The study is a randomised, double-blind, placebo-controlled, 3-period crossover, preceded by an open-label active-control period before randomisation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years-old.
* 18 ≤ BMI <30 kg/m².
* Clinical history consistent asthma, in the judgement of the investigator.
* Asthma controlled or partly controlled according to GINA 2012 criteria:
* Asthma treated by ICS and LABA (fixed-dose combination or free combination) at stable dose for at least 3 months.
* Able to replace the usual ICS and LABA therapy by ICS at the usual dose regimen and salbutamol as needed.
* Able to stop salbutamol at least 6 hours before a study visit.
* Able to perform at least 3 acceptable and reproducible FEV1 and FVC measurements according to ERS/ATS 2005 recommendations.

Exclusion Criteria:

* Clinically significant respiratory conditions other than asthma (e.g. pneumonia, pneumothorax, atelectasis, bronchiectasis, chronic bronchitis, COPD, emphysema, pulmonary arterial hypertension, pulmonary fibrosis,etc.).
* Upper or lower respiratory tract infection within 4 weeks.
* Exacerbation (requiring oral corticosteroids or hospitalization) within 3 months.
* Current smoker or former smoker less than 6 months or total lifetime smoking history greater than 10 pack-years.
* Intolerance to salbutamol.
* Intolerance to tiotropium (or any other atropine-derived compound).
* Intolerance to one of the ingredients of the study product
* Severe hepatic impairment, moderate to severe renal impairment, epilepsy, narrow angle glaucoma, gastrointestinal obstruction, moderate to severe prostatic hypertrophy, bladder neck obstruction.
* Any acute or chronic disease that will not allow the participation in the study, in the judgement of the investigator.
* Clinically relevant physical examination abnormality.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Normalised AUC 0-24h of FEV1 at day 8 of treatment period | At the 8th day of treatment period
  FEV1 assessed by spirometry

SECONDARY OUTCOMES:
Parameters of the pulmonary function | Day 1 and Day 8 of treatment period
  as well as the following criteria assessed the first day and the last day of each treatment period and the difference between the last day and the first day within each treatment periodadjusted for placebo effect:
  * the normalised AUC0-9h of FEV1 (L),
  * the normalised AUC0-12h of FEV1 (L),
  * the peak of FEV1 (L) which is the higher observed post-dosing value,
  * the trough of FEV1 (L) which is the last measurement before the next dosing (i.e. t24h),
  * the normalised AUC0-9h,AUC0-12h, AUC0-24h, peak and trough of FVC, MEF25, MEF50, MEF75, and MEF25-75.
PEF | Morning and evening from Day 1 to day 8 of treatment period
  PEF measured using a peak-flow meter
Dyspnoea | Day 1 to Day 8 of treatment period
  The criteria will be the normalised AUC0-9h,AUC0-12h, and AUC0-24h of the dyspnoea measurements(mm) assessed the first and the last day of each treatment period, and the difference between the last and the first day within each treatment period.
Vital signs | Visit 2, and at Visit 3 to Visit 10 (within 30 min pre-dose and 15 min, 30 min, 1 h, 2 h, 4 h, 6 h, 8 h, 24 h post-dose during the in-clinic visits) and at Visit 11
12-lead standard ECG | at Visit 1, at Visit 3 to Visit 10 (within 30 min pre-dose and 15 min, 1 h, 6 h, 24 h post-dose) and at Visit 11
Holter-ECG | At Visit 3 to Visit 10 : from 30 min pre-dose to 12 hours post-dose
Clinical laboratory tests (haematology, biochemistry, urinalysis) | Visit 1 and Visit 11
AEs | From Visit 1 to Visit 11
Normalised AUC 0-24h of FEV1 at Day 1 of treatment period | The first day of treatment period
  FEV1 assessed by spirometry
Difference between day 8 and first day of treatment period in normalised AUC 0-24h of FEV1 | Difference between day 8 and first day of treatement period
  FEV1 assessed by spirometry

CONTACTS AND LOCATIONS:
Locations (1):
- CRO, Gauting, Germany